CLINICAL TRIAL: NCT06156046
Title: Elucidation of the Mechanism of Immune Tolerance in Beekeepers
Brief Title: Tolerance in Beekeepers
Status: Recruiting | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor
Other Study IDs: 330722
Record Dates: First submitted 2023-11-24; First posted 2023-12-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Bee Sting
Keywords: Immune tolerance; Anaphylaxis; Beekeepers
MeSH Terms: conditions — Anaphylaxis | interventions — Patch Tests; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood-EDTA (Serum, PBMCs, Buffy coats, DNA & RNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Individuals naïve to beekeeping (<2 previous bee stings, non in the last 24 months). No history of anaphylaxis
  Interventions: Diagnostic Test: skin prick test; Diagnostic Test: Blood tests
- Group 2: Beekeepers with > approximately 10 stings/year who have been beekeeping for >3 years. No history of anaphylaxis.
  Interventions: Diagnostic Test: skin prick test; Diagnostic Test: Blood tests
- Group 3: Beekeepers with diagnosis of anaphylaxis to bee venom in the last 12 months who are sensitised to bee venom ( as evidenced by positive IgE and positive skin test to bee venom)
  Interventions: Diagnostic Test: skin prick test; Diagnostic Test: Blood tests

INTERVENTIONS:
Diagnostic Test: skin prick test — Skin prick test for bee venom
Diagnostic Test: Blood tests — IgE/G and T cell tolerance studies

SUMMARY:
Beekeepers experience multiple bee stings each year. Many of these beekeepers (25-60%) become sensitized to bee venom through the production of specific antibodies that target the bee venom. Although these antibodies are important in the triggering of an allergic reaction only a small number of sensitised beekeepers go on to have an allergic reaction with symptoms away from the site of the sting. These reactions can be severe and are known as anaphylactic reactions.

The study investigates why some beekeepers develop severe allergic symptoms after bee stings while others do not.

This study will explore factors in the blood that protect sensitised individuals from having anaphylactic reactions - meaning that despite being sensitised they are tolerant and do not react to subsequent stings.

DETAILED DESCRIPTION:
Beekeepers experience multiple stings each year many of whom (25-60%) become sensitised to bee (apis mellifera) venom through the production of IgE antibodies. However only a small proportion of the sensitised group go on to have anaphylaxis to bee venom. This study will investigate differences in T cell tolerance to bee venom in 3 groups by exploring factors that "protect" sensitised individuals from having anaphylactic reactions - meaning that despite being sensitised they are tolerant and do not react to subsequent stings.

T regulatory cell (Tregs) play a critical role in promoting immune tolerance to allergens and Treg generation has been shown to occur in bee venom allergic individuals following venom desensitisation therapy. Observations in sensitised tolerant (non-allergic) beekeepers (TB) suggest that exposure to venom through bee stings results in a similar increase in the frequencies of induced Tregs (iTregs). Helios negative induced Treg cells have also been suggested to contribute significantly to the establishment of immune tolerance in beekeepers. We will analyse the differences in Treg and Teffector (Teff) populations comparing sensitised beekeepers who are able to tolerate venom exposure (sensitised, tolerant beekeepers TB) with those beekeepers who do develop symptoms of systemic allergic reactions following bee sting (AB). A group of non-sensitised (NS) individuals will be recruited as a control population. We will perform RNA-seq to analyse the gene expression in Treg cells and Teff cells from all three groups. This will help to identify molecular targets that are involved in inducing the allergic reaction and also the genes that are involved in suppressing this reaction.

Considering the outcome of tolerance or anaphylaxis following bee stings, and the role of Treg and Teff cells in these processes, we will investigate the epigenetic regulations involved, which determine these cell's function. RNA-seq analysis will provide critical information about the genes involved in allergic reaction or in its suppression. DNA and histone modification analyses in the regulatory regions of these genes will help to better understand the underlying mechanism.

This project will investigate why some beekeepers who are sensitised to bee venom are able to tolerate bee stings, while in other sensitised individuals a bee sting can lead to life threatening anaphylaxis. This is not only of significance to beekeepers, but also has potential implications for the understanding of allergen tolerance in other allergic disease.

ELIGIBILITY:
Inclusion Criteria:

- Group 1 inclusion criteria.

* Individuals naive to beekeeping (<2 previous bee stings, none in the last 24 months)
* no history of anaphylaxis to stings. Group 2 inclusion criteria.
* Beekeepers with > approximately 10 stings/year who have been beekeeping for >3 years.
* No history of anaphylaxis to bee venom. Group 3 inclusion criteria
* Beekeepers with diagnosis of anaphylaxis to bee venom in the last 12 months who are sensitised to bee venom (as evidenced by positive specific IgE and positive skin test to bee venom)

Exclusion Criteria:

* Unable to understand protocol/consent.
* Unable to commit to follow up visits.
* Participants with a known history of mastocytosis or under investigation for suspected mastocytosis.
* Participants undergoing desensitisation treatment to bee venom before the first visit.
* Participants being treatment with immunosuppressive medications. being treatment with immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 inclusion criteria. Individuals naive to beekeeping (<2 previous bee stings, none in the last 24 months).
  No history of anaphylaxis to bee stings.
  Group 2 inclusion criteria. Beekeepers with > approximately 10 stings/year who have been beekeeping for >3 years.
  No history of anaphylaxis to bee stings.
  Group 3 inclusion criteria Beekeepers with diagnosis of anaphylaxis to bee venom in the last 12 months who are sensitised to bee venom (as evidenced by positive specific IgE and positive skin test to bee venom).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Cell comparison | 3 years
  (i) To compare the number of various cell (CD4+, CD8+ and Treg etc.) populations in the non-sensitised control population (NS), the sensitised but tolerant beekeepers (TB) and the allergic beekeeper (AB) population.
Cellular function | 3 years
  (ii) To identify differences in cellular function in the non-sensitised control population (NS), the sensitised but tolerant beekeepers (TB) and the allergic beekeeper (AB) population.
Molecular mechanism | 3 years
  (iii) To elucidate the molecular mechanism and the differences observed in (i) and (ii).
Epi regulation | 3 years
  (iiii) To elucidate the epigenetic regulation underpinning and the differences observed in (i) and (ii)

SECONDARY OUTCOMES:
Sensitisation data- skin prick testing | 3 years
  To compare results of skin prick testing from the beginning and end of the beekeeping season.
Sensitisation data - specific IgE's in blood | 3 years
  To compare results of specific IgE's in blood from the beginning and end of the beekeeping season.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Bethune, Principal Investigator — University Hospitals Plymouth
Locations (1):
- Derriford Hospital - University Hospitals Plymouth, Plymouth, Devon, United Kingdom